CLINICAL TRIAL: NCT00874731
Title: A Clinical Trial to Assess the Effect of Ridaforolimus (AP23573; MK-8669) on QTc Interval in Patients
Brief Title: A Study to Evaluate the Effect of MK-8669 (Ridaforolimus) on QTc Interval in Participants With Advanced Cancer (MK-8669-037)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 8669-037; 2009_569 (Other: NIH); MK-8669-037 (Other: Merck Protocol Number)
Record Dates: First submitted 2009-03-31; First posted 2009-04-02 (Estimated); Results first posted 2019-05-06 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-04

CONDITIONS: Metastatic or Locally Advanced Cancer
MeSH Terms: conditions — Neoplasm Metastasis | interventions — ridaforolimus

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be blinded to treatment during Part 1 only.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pt 1. Placebo/Ridaforolimus 100 mg; Pt 2. Ridaforolimus 40 mg (Experimental): [Pt 1, Day 1]: Participants received a single dose of placebo (10 oral tablets) on Day 1 of Part 1. [Pt 1, Day 2]: Following completion of Part 1 / Day 1, participants received a single dose of ridaforolimus 100 mg (10 x 10 mg oral tablets) on Day 2 of Part 1. Following completion of Part 1 / Day 2, participants entered a washout period of ≥5 days before the first dose Part 2. [Pt 2]: Following completion of Part 1, participants received ridaforolimus 40 mg (4 x 10 mg oral tablets) given once daily (QD) for 5 consecutive days followed by 2 days off-drug.
  Interventions: Drug: Ridaforolimus 100 mg; Drug: Ridaforolimus 40 mg; Drug: Placebo

INTERVENTIONS:
Drug: Ridaforolimus 100 mg — Part 1: A single oral dose of 100 mg ridaforolimus (10 x 10 mg tablets) was given on Day 2.
  Other Names: AP23573; MK-8669; deforolimus (until May 2009)
Drug: Ridaforolimus 40 mg — Part 2 (optional): Ridaforolimus 40 mg (4 x 10 mg tablets) was received on a regimen of daily oral doses for 5 consecutive days followed by 2 days off-drug.
  Other Names: AP23573; MK-8669; deforolimus (until May 2009)
Drug: Placebo — Part 1: A single oral dose of placebo (10 x placebo tablets) was given on Day 1.

SUMMARY:
To assess the potential for ridaforolimus to prolong the QTc interval (an effect on the electrical activity of the heart) in participants with advanced cancer. This study will be done in 2 parts. Part 1 (Pt 1) will evaluate the effect of a single 100 mg dose of ridaforolimus on QT interval in participants with advanced cancer. Fridericias's correction (QTcF) will be used. In Part 2 (Pt 2), participants will receive ridaforolimus at the current therapeutic dose (40 mg x 5 days).

ELIGIBILITY:
Inclusion Criteria:

* Participant must have metastatic or locally advanced cancer which has failed to respond to standard therapy or no therapy exists.
* If the participant is a female, she must be postmenopausal or if she is of childbearing potential she must have blood pregnancy tests during the study and be willing to use 2 methods of contraception.
* If the participant is male and has female partners of child-bearing potential, he must agree to use a medically acceptable method of contraception during the study and for 30 days after the last dose of study drug.

Exclusion Criteria:

* Participant has had chemotherapy, radiotherapy or biological therapy within the past 4 weeks.
* Participant is currently receiving other anti-cancer therapy.
* Participant is currently participating or has participated in a study with an investigation drug or device within the last 30 days.
* Participant has a primary central nervous system tumor or active brain metastases.
* Participant has a psychiatric disorder.
* Participant uses illegal drugs.
* Participant is pregnant or breastfeeding.
* Participant is known to be human immunodeficiency virus (HIV) positive.
* Participant has a known history of Hepatitis B or C.
* Participant has newly diagnosed diabetes.
* Participant has an active infection.
* Participant is unable to swallow capsules.
* Participant has received a blood transfusion with one week of study entry.
* Participant has a history of cardiac problems including heart failure, myocardial infarction, unstable angina, congestive heart failure or cardiac arrhythmia.
* Participant has a known sensitivity to the components of the study drug.
* Participant has not adequately recovered from any prior surgical procedure.
* Participant does not agree to refrain from use of herbal remedies and consumption of grapefruit juice for 2 weeks prior to and during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-04-28 (Actual); Primary Completion 2009-10-30 (Actual); Study Completion 2010-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Lush RM, Patnaik A, Sullivan D, Papadopoulos KP, Trucksis M, McCrea J, Cerchio K, Li X, Stroh M, Selverian D, Orford K, Ebbinghaus S, Agrawal N, Iwamoto M, Wagner JA, Tolcher A. A single supratherapeutic dose of ridaforolimus does not prolong the QTc interval in patients with advanced cancer. Cancer Chemother Pharmacol. 2012 Oct;70(4):567-74. doi: 10.1007/s00280-012-1942-7. Epub 2012 Aug 10. PMID 22878520

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of N=23 participants were enrolled in this study, conducted in 2 parts. Participants completing study Part 1 (Pt 1) had the option to continue to Part 2 (Pt 2).
Pre-assignment Details: Participants progressed through the study as a single group over 4 periods: 1) Pt 1, Day 1: Placebo; 2) Pt 1, Day 2: Ridaforolimus 100 mg; 3) washout period (≥5 days); and 4) Part 2: Ridaforolimus 40 mg.
Groups:
- Pt 1, Day 1. Placebo: [Pt 1, Day 1]: Participants received a single dose of placebo (10 oral tablets) on Day 1 of Part 1.
- Pt 1, Day 2. Ridaforolimus 100 mg: [Pt 1, Day 2]: Following completion of Part 1 / Day 1, participants received a single dose of ridaforolimus 100 mg (10 x 10 mg oral tablets) on Day 2 of Part 1. Following completion of Part 1 / Day 2, participants entered a washout period of ≥5 days before the first dose Part 2.
- Pt 2. Ridaforolimus 40 mg: [Pt 2]: Following completion of Part 1, participants received ridaforolimus 40 mg (4 x 10 mg oral tablets) given once daily (QD) for 5 consecutive days followed by 2 days off-drug.
Period: Part 1, Day 1: Placebo
Arm/Group | Pt 1, Day 1. Placebo | Pt 1, Day 2. Ridaforolimus 100 mg | Pt 2. Ridaforolimus 40 mg
Started | 23 | 0 | 0
Completed | 22 | 0 | 0
Not Completed | 1 | 0 | 0
Not completed — Disease Progression | 1 | 0 | 0
Period: Part 1, Day 2: Ridaforolimus 100 mg
Arm/Group | Pt 1, Day 1. Placebo | Pt 1, Day 2. Ridaforolimus 100 mg | Pt 2. Ridaforolimus 40 mg
Started | 0 (Participants completing Pt 1, Day 1, enter into the "Pt 1, Day 2. Ridaforolimus 100 mg" arm.) | 22 (Participants completing Pt 1, Day 1, started this period in "Pt 1, Day 2. Ridaforolimus 100 mg" arm.) | 0
Completed | 0 | 22 | 0
Not Completed | 0 | 0 | 0
Period: Washout Period
Arm/Group | Pt 1, Day 1. Placebo | Pt 1, Day 2. Ridaforolimus 100 mg | Pt 2. Ridaforolimus 40 mg
Started | 0 | 22 | 0
Completed | 0 | 22 | 0
Not Completed | 0 | 0 | 0
Period: Part 2: Ridaforolimus 40 mg
Arm/Group | Pt 1, Day 1. Placebo | Pt 1, Day 2. Ridaforolimus 100 mg | Pt 2. Ridaforolimus 40 mg
Started | 0 | 0 (Participants completing Pt 1 and washout, enter into the "Pt 2. Ridaforolimus 40 mg" arm.) | 22 (Participants completing Pt 1 and washout, started this period in "Pt 2. Ridaforolimus 40 mg" arm.)
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 22
Not completed — Adverse Event | 0 | 0 | 3
Not completed — Disease Progression | 0 | 0 | 19

BASELINE CHARACTERISTICS:
Population: Baseline data are reported for all participants starting the study on Day 1 of Part 1, receiving placebo treatment.
Arm/Group | Pt 1, Day 1. Placebo
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (11.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Part 1. Mean Change From Baseline in Rate-Corrected (Fridericia's) QT Interval (QTcF) at 0.5 Hours
Description: The mean change from baseline (CFB) in QTcF at 0.5 hours post-dose was assessed. At baseline (pre-dose) and at 0.5 hours post-dose, 5 replicate electrocardiograms (ECGs) were collected to reduce measurement variability. The 5 replicate QTcF values were averaged to calculate the QTcF value for each participant. Further, each participant served as their own control for the calculation of CFB in QTcF after placebo and ridaforolimus 100 mg dosing. Additionally, CFB in QTcF after single ridaforolimus 100 mg dosing for each participant was adjusted for the CFB in QTcF observed after placebo dosing.
Time Frame: Baseline and 0.5 hours post-dose on Days 1 & 2 of Part 1
Population: Includes only participants in Part 1 receiving treatment. QTcF not analyzed in Part 2. QTcF data are excluded from: 1) both arms (N=1; non-evaluable ECG waveform); and 2) ridaforolimus arm (N=2; protocol violation & study discontinuation).
Measure: Mean (95% Confidence Interval); unit: milliseconds (msec)
Arm/Group | Pt 1, Day 1. Placebo | Pt 1, Day 2. Ridaforolimus 100 mg
Number analyzed (Participants) | 22 | 20
milliseconds (msec)
  Baseline (Pre-dose) | 419.23 [412.61 to 425.86] | 418.08 [411.40 to 424.75]
  Change from Baseline at 0.5 Hours | 1.42 [-1.89 to 4.74] | 1.90 [-1.53 to 5.33]
Statistical Analysis 1: Comparison: Pt 1, Day 1. Placebo vs Pt 1, Day 2. Ridaforolimus 100 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.48, 90% CI 2-sided [-2.80 to 3.76] — Mean Difference in CFB = Ridaforolimus - Placebo; Mean difference and 90% confidence interval generated using a repeated measures mixed model that included treatment, time and treatment-by-time interaction as fixed factors and subject as random factor

2. Secondary Outcome: Number of Participants Experiencing an Adverse Event (AE)
Description: The number of participants experiencing an AE was assessed. An AE was defined as any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE. Participants experiencing AEs were counted under the treatment they received when the AE occurred. Participants experiencing AEs during the washout period between Part 1 and Part 2 are counted in the "Pt 1, Day 2. Ridaforolimus 100 mg" arm.
Time Frame: Up to 7 months
Population: All participants receiving ≥1 dose of study treatment. The washout period following Part 1 was the safety follow-up period for Part 1. For this reason, AEs that occurred during the washout period are appropriately included as Part 1 AEs. One participant discontinued after the Day 1 placebo dose and did not receive ridaforolimus 100 mg or 40 mg.
Measure: Count of Participants; unit: Participants
Arm/Group | Pt 1, Day 1. Placebo | Pt 1, Day 2. Ridaforolimus 100 mg | Pt 2. Ridaforolimus 40 mg
Number analyzed (Participants) | 23 | 22 | 22
Participants | 11 | 18 | 21

3. Secondary Outcome: Number of Participants Discontinuing Study Treatment Due to an Adverse Event
Description: The number of participants discontinuing study treatment due to an AE was assessed. An AE was defined as any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE. Participants discontinuing study treatment due to an AE were counted as discontinuing under the treatment they received when the AE occurred.
Time Frame: Up to 6 months
Population: All participants receiving ≥1 dose of study treatment. One participant discontinued from study after the Day 1 placebo dose and did not receive ridaforolimus 100 mg or 40 mg.
Measure: Count of Participants; unit: Participants
Arm/Group | Pt 1, Day 1. Placebo | Pt 1, Day 2. Ridaforolimus 100 mg | Pt 2. Ridaforolimus 40 mg
Number analyzed (Participants) | 23 | 22 | 22
Participants | 0 | 0 | 3

4. Primary Outcome: Part 1. Mean Change From Baseline in Rate-Corrected (Fridericia's) QT Interval (QTcF) at 1 Hour
Description: The mean change from baseline (CFB) in QTcF at 1 hour post-dose was assessed. At baseline (pre-dose) and at 1 hour post-dose, 5 replicate electrocardiograms (ECGs) were collected to reduce measurement variability. The 5 replicate QTcF values were averaged to calculate the QTcF value for each participant. Further, each participant served as their own control for the calculation of CFB in QTcF after placebo and ridaforolimus 100 mg dosing. Additionally, CFB in QTcF after single ridaforolimus 100 mg dosing for each participant was adjusted for the CFB in QTcF observed after placebo dosing.
Time Frame: Baseline and 1 hour post-dose on Days 1 & 2 of Part 1
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: msec
Arm/Group | Pt 1, Day 1. Placebo | Pt 1, Day 2. Ridaforolimus 100 mg
Number analyzed (Participants) | 22 | 20
msec
  Baseline (Pre-dose) | 419.23 [412.61 to 425.86] | 418.08 [411.40 to 424.75]
  Change from Baseline at 1 Hour | 2.40 [-0.92 to 5.71] | 1.85 [-1.58 to 5.28]
Statistical Analysis 1: Comparison: Pt 1, Day 1. Placebo vs Pt 1, Day 2. Ridaforolimus 100 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.54, 95% CI 2-sided [-3.83 to 2.74] — Mean Difference in CFB = Ridaforolimus - Placebo; [other analysis details as in outcome 1, analysis 1]

5. Primary Outcome: Part 1. Mean Change From Baseline in Rate-Corrected (Fridericia's) QT Interval (QTcF) at 2 Hours
Description: The mean change from baseline (CFB) in QTcF at 2 hours post-dose was assessed. At baseline (pre-dose) and at 2 hours post-dose, 5 replicate electrocardiograms (ECGs) were collected to reduce measurement variability. The 5 replicate QTcF values were averaged to calculate the QTcF value for each participant. Further, each participant served as their own control for the calculation of CFB in QTcF after placebo and ridaforolimus 100 mg dosing. Additionally, CFB in QTcF after single ridaforolimus 100 mg dosing for each participant was adjusted for the CFB in QTcF observed after placebo dosing.
Time Frame: Baseline and 2 hours post-dose on Days 1 & 2 of Part 1
Population: Includes only participants in Part 1 receiving treatment. QTcF not analyzed in Part 2. QTcF data are excluded from: 1) both arms (N=1; non-evaluable ECG waveform); and 2) ridaforolimus arm (N=2; protocol violation & study discontinuation). Further, CFB data are excluded from the placebo arm for missing data (N=1).
Measure: Mean (95% Confidence Interval); unit: msec
Arm/Group | Pt 1, Day 1. Placebo | Pt 1, Day 2. Ridaforolimus 100 mg
Number analyzed (Participants) | 22 | 20
msec
  Baseline (Pre-dose) | 419.23 [412.61 to 425.86] | 418.08 [411.40 to 424.75]
  Change from Baseline at 2 Hours: number analyzed (Participants) | 21 | 20
  Change from Baseline at 2 Hours | 2.40 [-0.97 to 5.77] | 1.22 [-2.21 to 4.65]
Statistical Analysis 1: Comparison: Pt 1, Day 1. Placebo vs Pt 1, Day 2. Ridaforolimus 100 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -1.18, 95% CI 2-sided [-4.50 to 2.14] — Mean Difference in CFB = Ridaforolimus - Placebo; [other analysis details as in outcome 1, analysis 1]

6. Primary Outcome: Part 1. Mean Change From Baseline in Rate-Corrected (Fridericia's) QT Interval (QTcF) at 3 Hours
Description: The mean change from baseline (CFB) in QTcF at 3 hours post-dose was assessed. At baseline (pre-dose) and at 3 hours post-dose, 5 replicate electrocardiograms (ECGs) were collected to reduce measurement variability. The 5 replicate QTcF values were averaged to calculate the QTcF value for each participant. Further, each participant served as their own control for the calculation of CFB in QTcF after placebo and ridaforolimus 100 mg dosing. Additionally, CFB in QTcF after single ridaforolimus 100 mg dosing for each participant was adjusted for the CFB in QTcF observed after placebo dosing.
Time Frame: Baseline and 3 hours post-dose on Days 1 & 2 of Part 1
Population: as for outcome 5
Measure: Mean (95% Confidence Interval); unit: msec
Arm/Group | Pt 1, Day 1. Placebo | Pt 1, Day 2. Ridaforolimus 100 mg
Number analyzed (Participants) | 22 | 20
msec
  Baseline (Pre-dose) | 419.23 [412.61 to 425.86] | 418.08 [411.40 to 424.75]
  Change from Baseline at 3 Hours: number analyzed (Participants) | 21 | 20
  Change from Baseline at 3 Hours | 2.94 [-0.42 to 6.31] | 3.41 [-0.02 to 6.84]
Statistical Analysis 1: Comparison: Pt 1, Day 1. Placebo vs Pt 1, Day 2. Ridaforolimus 100 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.47, 95% CI 2-sided [-2.85 to 3.79] — Mean Difference in CFB = Ridaforolimus - Placebo; [other analysis details as in outcome 1, analysis 1]

7. Primary Outcome: Part 1. Mean Change From Baseline in Rate-Corrected (Fridericia's) QT Interval (QTcF) at 4 Hours
Description: The mean change from baseline (CFB) in QTcF at 4 hours post-dose was assessed. At baseline (pre-dose) and at 4 hours post-dose, 5 replicate electrocardiograms (ECGs) were collected to reduce measurement variability. The 5 replicate QTcF values were averaged to calculate the QTcF value for each participant. Further, each participant served as their own control for the calculation of CFB in QTcF after placebo and ridaforolimus 100 mg dosing. Additionally, CFB in QTcF after single ridaforolimus 100 mg dosing for each participant was adjusted for the CFB in QTcF observed after placebo dosing.
Time Frame: Baseline and 4 hours post-dose on Days 1 & 2 of Part 1
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: msec
Arm/Group | Pt 1, Day 1. Placebo | Pt 1, Day 2. Ridaforolimus 100 mg
Number analyzed (Participants) | 22 | 20
msec
  Baseline (Pre-dose) | 419.23 [412.61 to 425.86] | 418.08 [411.40 to 424.75]
  Change from Baseline at 4 Hours | 1.32 [-1.99 to 4.64] | 2.51 [-0.92 to 5.94]
Statistical Analysis 1: Comparison: Pt 1, Day 1. Placebo vs Pt 1, Day 2. Ridaforolimus 100 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 1.18, 95% CI 2-sided [-2.10 to 4.47] — Mean Difference in CFB = Ridaforolimus - Placebo; [other analysis details as in outcome 1, analysis 1]

8. Primary Outcome: Part 1. Mean Change From Baseline in Rate-Corrected (Fridericia's) QT Interval (QTcF) at 6 Hours
Description: The mean change from baseline (CFB) in QTcF at 6 hours post-dose was assessed. At baseline (pre-dose) and at 6 hours post-dose, 5 replicate electrocardiograms (ECGs) were collected to reduce measurement variability. The 5 replicate QTcF values were averaged to calculate the QTcF value for each participant. Further, each participant served as their own control for the calculation of CFB in QTcF after placebo and ridaforolimus 100 mg dosing. Additionally, CFB in QTcF after single ridaforolimus 100 mg dosing for each participant was adjusted for the CFB in QTcF observed after placebo dosing.
Time Frame: Baseline and 6 hours post-dose on Days 1 & 2 of Part 1
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: msec
Arm/Group | Pt 1, Day 1. Placebo | Pt 1, Day 2. Ridaforolimus 100 mg
Number analyzed (Participants) | 22 | 20
msec
  Baseline (Pre-dose) | 419.23 [412.61 to 425.86] | 418.08 [411.40 to 424.75]
  Change from Baseline at 6 Hours | -3.37 [-6.68 to -0.06] | -0.87 [-4.30 to 2.56]
Statistical Analysis 1: Comparison: Pt 1, Day 1. Placebo vs Pt 1, Day 2. Ridaforolimus 100 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 2.49, 95% CI 2-sided [-0.79 to 5.78] — Mean Difference in CFB = Ridaforolimus - Placebo; [other analysis details as in outcome 1, analysis 1]

9. Primary Outcome: Part 1. Mean Change From Baseline in Rate-Corrected (Fridericia's) QT Interval (QTcF) at 8 Hours
Description: The mean change from baseline (CFB) in QTcF at 8 hours post-dose was assessed. At baseline (pre-dose) and at 8 hours post-dose, 5 replicate electrocardiograms (ECGs) were collected to reduce measurement variability. The 5 replicate QTcF values were averaged to calculate the QTcF value for each participant. Further, each participant served as their own control for the calculation of CFB in QTcF after placebo and ridaforolimus 100 mg dosing. Additionally, CFB in QTcF after single ridaforolimus 100 mg dosing for each participant was adjusted for the CFB in QTcF observed after placebo dosing.
Time Frame: Baseline and 8 hours post-dose on Days 1 & 2 of Part 1
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: msec
Arm/Group | Pt 1, Day 1. Placebo | Pt 1, Day 2. Ridaforolimus 100 mg
Number analyzed (Participants) | 22 | 20
msec
  Baseline | 419.23 [412.61 to 425.86] | 418.08 [411.40 to 424.75]
  Change from Baseline at 8 Hours | -5.27 [-8.58 to -1.96] | -2.79 [-6.22 to 0.64]
Statistical Analysis 1: Comparison: Pt 1, Day 1. Placebo vs Pt 1, Day 2. Ridaforolimus 100 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 2.48, 95% CI 2-sided [-0.80 to 5.76] — Mean Difference in CFB = Ridaforolimus - Placebo; [other analysis details as in outcome 1, analysis 1]

10. Primary Outcome: Part 1. Mean Change From Baseline in Rate-Corrected (Fridericia's) QT Interval (QTcF) at 10 Hours
Description: The mean change from baseline (CFB) in QTcF at 10 hours post-dose was assessed. At baseline (pre-dose) and at 10 hours post-dose, 5 replicate electrocardiograms (ECGs) were collected to reduce measurement variability. The 5 replicate QTcF values were averaged to calculate the QTcF value for each participant. Further, each participant served as their own control for the calculation of CFB in QTcF after placebo and ridaforolimus 100 mg dosing. Additionally, CFB in QTcF after single ridaforolimus 100 mg dosing for each participant was adjusted for the CFB in QTcF observed after placebo dosing.
Time Frame: Baseline and 10 hours post-dose on Days 1 & 2 of Part 1
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: msec
Arm/Group | Pt 1, Day 1. Placebo | Pt 1, Day 2. Ridaforolimus 100 mg
Number analyzed (Participants) | 22 | 20
msec
  Baseline (Pre-dose) | 419.23 [412.61 to 425.86] | 418.08 [411.40 to 424.75]
  Change from Baseline at 10 Hours | -5.00 [-8.32 to -1.69] | -1.12 [-4.55 to 2.31]
Statistical Analysis 1: Comparison: Pt 1, Day 1. Placebo vs Pt 1, Day 2. Ridaforolimus 100 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 3.89, 95% CI 2-sided [0.60 to 7.17] — Mean Difference in CFB = Ridaforolimus - Placebo; [other analysis details as in outcome 1, analysis 1]

11. Primary Outcome: Part 1. Mean Change From Baseline in Rate-Corrected (Fridericia's) QT Interval (QTcF) at 24 Hours
Description: The mean change from baseline (CFB) in QTcF at 24 hours post-dose was assessed. At baseline (pre-dose) and at 24 hours post-dose, 5 replicate electrocardiograms (ECGs) were collected to reduce measurement variability. The 5 replicate QTcF values were averaged to calculate the QTcF value for each participant. Further, each participant served as their own control for the calculation of CFB in QTcF after placebo and ridaforolimus 100 mg dosing. Additionally, CFB in QTcF after single ridaforolimus 100 mg dosing for each participant was adjusted for the CFB in QTcF observed after placebo dosing.
Time Frame: Baseline and 24 hours post-dose on Days 1 & 2 of Part 1
Population: Includes only participants in Part 1 receiving treatment. QTcF not analyzed in Part 2. QTcF data are excluded from: 1) both arms (N=1; non-evaluable ECG waveform); and 2) ridaforolimus arm (N=2; protocol violation & study discontinuation). Further, CFB data are excluded from the placebo arm for missing data (N=1) and study discontinuation (N=1).
Measure: Mean (95% Confidence Interval); unit: msec
Arm/Group | Pt 1, Day 1. Placebo | Pt 1, Day 2. Ridaforolimus 100 mg
Number analyzed (Participants) | 22 | 20
msec
  Baseline (Pre-dose) | 419.23 [412.61 to 425.86] | 418.08 [411.40 to 424.75]
  Change from Baseline at 24 Hours: number analyzed (Participants) | 20 | 20
  Change from Baseline at 24 Hours | -0.74 [-4.17 to 2.69] | -2.24 [-5.67 to 1.19]
Statistical Analysis 1: Comparison: Pt 1, Day 1. Placebo vs Pt 1, Day 2. Ridaforolimus 100 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -1.50, 95% CI 2-sided [-4.85 to 1.86] — Mean Difference in CFB = Ridaforolimus - Placebo; [other analysis details as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Up to 7 months
Description: The analysis population included all participants receiving ≥1 dose of study treatment. Participants with adverse events (AEs) were counted under the treatment received when the AE occurred. AEs that occurred during the washout period between Part 1 and Part 2 are counted in the "Pt 1, Day 2. Ridaforolimus 100 mg" arm. The washout period following Part 1 was the safety follow-up period for Part 1 and AEs that occurred during the washout period are appropriately included as Part 1 AEs.
Arm/Group | Pt 1, Day 1. Placebo | Pt 1, Day 2. Ridaforolimus 100 mg | Pt 2. Ridaforolimus 40 mg
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/22 | 2/22
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/22 | 8/22
Other Adverse Events (participants affected / at risk) | 8/23 | 18/22 | 21/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pt 1, Day 1. Placebo (N=23) | Pt 1, Day 2. Ridaforolimus 100 mg (N=22) | Pt 2. Ridaforolimus 40 mg (N=22)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchitis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vulval abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pt 1, Day 1. Placebo (N=23) | Pt 1, Day 2. Ridaforolimus 100 mg (N=22) | Pt 2. Ridaforolimus 40 mg (N=22)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 4 (4) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2) | 4 (4) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 5 (5) | 4 (5)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 8 (8)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 3 (3)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 4 (4) | 6 (6)
Oedema (General disorders) | 0 (0) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 2 (2)
Fatigue (General disorders) | 0 (0) | 6 (6) | 9 (12)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 9 (10)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 3 (3)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Blood magnesium decreased (Investigations) | 3 (3) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 5 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (2)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) | 4 (5)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3)
Haematuria (Renal and urinary disorders) | 1 (1) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 4 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication guidelines.